CLINICAL TRIAL: NCT02508129
Title: Pragmatic Trial of Behavioral Interventions for Insomnia in Hypertensive Patients
Brief Title: Hypertension With Unsatisfactory Sleep Health
Acronym: HUSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Virginia (Other); Carolinas Medical Center (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Daniel J. Buysse, M.D., Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO14070337; UH2HL125103 (NIH)
Record Dates: First submitted 2015-07-21; First posted 2015-07-24 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Insomnia; Hypertension
Keywords: Insomnia; hypertension; blood pressure; sleep; behavioral treatment; Cognitive Behavioral Treatment of Insomnia (CBTI); Brief Behavioral Treatment of Insomnia (BBTI); pragmatic trial; internet
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Brief Behavioral Treatment for Insomnia (Experimental): Brief Behavioral Treatment for Insomnia (BBTI) employs behavioral strategies for managing insomnia and is administered in 4 brief weekly contacts with a therapist via online web conferencing.
  Interventions: Behavioral: Brief Behavioral Treatment for Insomnia
- Sleep Healthy Using the Internet (SHUTi) (Experimental): SHUTi is an automated, interactive, personalized web-based program for improving insomnia through the use of Cognitive-Behavioral Therapy strategies for insomnia.
  Interventions: Behavioral: Sleep Healthy Using the Internet
- Enhanced Usual Care (EUC) (Placebo Comparator): EUC involves the primary care physician's current treatment; feedback to patients and providers on assessment and treatment recommendations; an educational video from Emmi Solutions, Inc.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Brief Behavioral Treatment for Insomnia — BBTI employs behavioral strategies for treating insomnia, including stimulus control and sleep restriction. The BBTI interventionist contacts occur by telephone or web conferencing. It is administered in an initial session, followed by 3 brief weekly contacts, each guided by a printed workbook. During an initial 60 minute session, the sleep interventionist will review the participant's insomnia symptoms, discuss sleep regulation, and develop an individualized prescription of sleep wake times.
  Other Names: BBTI
  Arms: Brief Behavioral Treatment for Insomnia
Behavioral: Sleep Healthy Using the Internet — SHUTi is a self-guided, automated, interactive, and tailored web-based program modeled on the primary tenets of Cognitive Behavioral Treatment for Insomnia (CBT-I): sleep restriction, stimulus control, cognitive restructuring, sleep hygiene, and relapse prevention. Intervention content is metered out over 6 Cores based on a time and event-based schedule. SHUTi uses online sleep diaries to track progress and to tailor treatment (e.g., assign a "sleep restriction" window). Each Core acts as an online analog for the weekly sessions of traditional CBT-I and follows the same structure.
  Other Names: SHUTi
  Arms: Sleep Healthy Using the Internet (SHUTi)
Behavioral: Enhanced Usual Care — Participants randomized to EUC will complete the standard panel of self-report assessments and home blood pressure monitoring at baseline. The study team will generate an individualized report based, which will be sent to the participant and physician. The report will also contain publically-available educational resources (websites, books) and contact information for treatment resources. Participants in EUC will be given a link to a website containing an educational video on insomnia and its treatment, produced by Emmi Solutions, Inc. Participants in EUC will complete outcome assessments on the same schedule as participants in the other conditions. Participants who complete the EUC intervention will be offered the CBT-I/ SHUTi intervention following study completion.
  Other Names: EUC
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
Insomnia and hypertension are common health problems that often occur together and influence each other. This practical, low-cost, clinical trial will evaluate two behavioral treatments for insomnia (a brief intervention with therapist contact and a self-guided Internet intervention) compared to usual care. Participants will be recruited using the electronic health record in their primary care physicians' offices, and will be evaluated for sleep, blood pressure, and health outcomes after 9 weeks, 6 months, and 12 months.

DETAILED DESCRIPTION:
Insomnia is a prevalent, chronic, and inadequately-treated chronic medical condition associated with comorbid conditions such as hypertension (HTN) and a range of adverse health outcomes. Hypnotic medications are efficacious and widely available, but they have potentially serious adverse effects. Patients and providers prefer non-drug treatments such as Cognitive-Behavioral Treatment of Insomnia (CBT-I), which is safe, efficacious, and durable-but not widely available. Innovative use of electronic health records (EHR) to identify patients, and the availability of new technologies that enable cognitive-behavioral interventions to be delivered at scale, with high treatment fidelity, and at low cost, offer exciting opportunities to address these critical problems. The investigators propose a low-cost, pragmatic, patient-centered, randomized controlled trial comparing two CBT-I-based interventions for insomnia with comorbid hypertension (INS+HTN) to primary care physicians' (PCP) enhanced usual care (EUC). The setting will be University of Pittsburgh Medical Center (UPMC) primary care practices. Participants will be 625 adults with INS+HTN. Recruitment will be conducted using alerts in the EpicCare EHR triggered by patient characteristics (hypertension; hypnotic medications or insomnia diagnosis/problem). The investigators will compare 3 interventions: Brief Behavioral Treatment of Insomnia (BBTI), involving electronic educational material and 4 telephone/web sessions with a live interventionist; "Sleep Healthy Using The Internet" (SHUTi), a self-guided, 8-module, Internet version of CBT-I, with no human contact; and EUC, which includes assessment and educational information for participants and providers. The primary outcome will be self-reported sleep at 9 weeks. Other outcomes include domains of symptoms, health, and patient/provider satisfaction obtained by self-report, home blood pressure monitoring (HBPM), and EHR. Specific Aims for the trial are: (1) To compare interventions on patient-reported symptoms at 9 weeks, 6 months, and 12 months. (2) To compare interventions on health indicators including self-report, HBPM, and EHR measures at 6 and 12 months. (3) To compare patient and provider-level satisfaction with the 3 interventions. (4) Exploratory Aim: To compare BBTI and CBT-I on each outcome domain and intervention adherence/drop-outs.

We made changes to the outcome measures document in April, 2019, and further amended these measures in June, 2019. The reason for these changes was to ensure consistency among the grant application, clinical trial protocol paper, and ClinicalTrials.gov. We made the following specific changes and corrections:

* Insomnia diagnosis, cumulative illness rating scale, and treatment expectations were removed as secondary outcomes, as they are not listed in our protocol as outcome measures. They are only measured at baseline to characterize participants.
* Health-Related Quality of Life "Medical Outcomes Survey Short Form-12 and Client Satisfaction "Client Satisfaction Questionnaire" were changed from primary to secondary outcome measures, to ensure consistency with the grant application and protocol paper.
* Side effects "Treatment-related Side Effects Scale" were changed from a secondary to an "other" outcome measure, again to ensure consistency with the grant application and protocol paper.

The following outcome measures were added to ClinicalTrials.gov to ensure consistency:

Secondary Outcome: Provider Satisfaction "Provider Satisfaction Survey"

Other Prespecified Outcome Measures:

* Daytime Impairment Related to Sleep "PROMIS Sleep Related Impairment"
* Insomnia Severity "Insomnia Severity Index"
* Sleep Quality "Pittsburgh Sleep Quality Index"
* Daytime Sleepiness "Epworth Sleepiness Scale"
* Falls "Side Effect/Falls Questionnaire" "Falls Follow-up Questionnaire"
* Improvement "Patient Global Impression of Improvement Scale"
* Sleep Diary Measures "HUSH Daily Diary"

We also recognized that we had erroneously interpreted "time frame" as the time frame of the instrument itself, rather than the time frame of the assessment battery. Time frames in ClinicalTrials.gov were corrected to capture the time points at which they are assessed, in the following measures:

* Sleep disturbance "PROMIS Sleep Disturbance Scale"
* Health related quality of life "Medical Outcomes Survey Short Form-12"
* Client satisfaction "Client Satisfaction Questionnaire"
* Depression "PROMIS Depression Scale"
* Anxiety "PROMIS Anxiety Scale"
* Fatigue "PROMIS Fatigue Scale"
* Blood pressure "HUSH Sleep Diary"
* Hypnotic use "Health Care Utilization Questionnaire" "HUSH Sleep Diary"
* Health care costs "Health Care Utilization Questionnaire"
* Side effects "Treatment-related Side Effects Scale"

ELIGIBILITY:
Inclusion Criteria:

1. Hypertension diagnosis 'Hypertension diagnosis' is indicated by the presence of at least one of the following:

   1. International Classification of Diseases, Ninth Revision, Clinical Modification (ICD-9-CM) diagnosis of essential hypertension in the electronic health record;
   2. Hypertension listed in the medical problem list in the electronic health record.
2. At least one of the following:

   1. Hypnotic on active med list
   2. Insomnia on diagnosis or problem list
3. Age 18 years and up.
4. Meets criteria for DSM-5 (Diagnostic and Statistical Manual of Mental Disorders-5th ed.) Insomnia Disorder
5. At least moderate insomnia severity: Score > 7 on Insomnia Severity Index
6. Telephone, e-mail address, reliable Internet access. 'Reliable internet access' is defined by an individual having a personal e-mail address and having regular internet access within his/her own residence.
7. Stable medical, psychiatric condition

Exclusion Criteria:

1. Untreated current major depression (Patient Health Questionnaire (PHQ-9) score equal to or greater than 15; Generalized Anxiety Disorder (GAD-7) score > 10); patients using stable (3 mos) medication, psychological treatment ARE eligible
2. History of bipolar disorder or psychosis
3. Substance use disorder within past 3 months
4. Dementia or probable dementia diagnosis
5. Active suicidal ideation or psychosis
6. Delayed sleep phase disorder (DSPD) or severe, untreated restless legs syndrome (RLS)
7. Plans to leave present source of care during the following year
8. Non-English speaking, illiterate, or sensory deficits
9. Shift work that includes working the night shift (between the hours of 12:00 a.m. - 6:00 a.m.)
10. Apnea Hypopnea Index (AHI) greater than or equal to 50 or O2 saturation 85% or less for > or = to 10% of the night.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2015-08; Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Sleep Disturbance | 9 weeks
  Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance:
  PROMIS Sleep Disturbance measures self-reported sleep quality and associated daytime functioning during the past seven days. It is administered by computerized adaptive testing (CAT) with individual responses guiding the system's choice of subsequent items from the full 27-item item bank.
  Scale Range: Item responses are combined to yield a T-score with population mean of 50, standard deviation of 10, and range of ~20 - ~80. Higher scores indicate greater Sleep Disturbance.

SECONDARY OUTCOMES:
Depression | 9 weeks, 6 months, 12 months
  The PROMIS Depression Scale is a self-report measure that assesses negative mood, views of self, social cognition, affect and engagement during the past seven days. It is administered by computerized adaptive testing (CAT) with individual responses guiding the system's choice of subsequent items from the full 28-item bank.
  Scale Range: Item responses are combined to yield a T-score with population mean of 50, standard deviation of 10, and range of ~20 - ~80. Higher scores indicate greater Depression.
Anxiety | 9 weeks, 6 months, 12 months
  The PROMIS Anxiety Scale is a self-report measure that assesses fear, anxiousness, and hyperarousal and its associated somatic symptoms during the past seven days. It is administered by computerized adaptive testing (CAT) with individual responses guiding the system's choice of subsequent items from the full 29-item bank.
  Scale Range: Item responses are combined to yield a T-score with population mean of 50, standard deviation of 10, and range of ~20 - ~80. Higher scores indicate greater Anxiety.
Fatigue | 9 weeks, 6 months, 12 months
  The PROMIS Fatigue Scale is a self-report measure that assesses the experience and impact of fatigue during the past seven days. It is administered by computerized adaptive testing (CAT) with individual responses guiding the system's choice of subsequent items from the full 95-item bank.
  Scale Range: Item responses are combined to yield a T-score with population mean of 50, standard deviation of 10, and range of ~20 - ~80. Higher scores indicate greater Fatigue.
Blood Pressure | 9 weeks, 6 months, 12 months
  Home blood pressures are measured with an Omron BP786 home blood pressure monitor. Reported values for each day in each participant represent the average systolic and diastolic readings and heart rate from 3 measurements. Participants record these values in a 7-day sleep diary. Daily measurements for each participant are averaged across the number of days of recording.
  Scale Range: Systolic BP range: 0 - 299; Diastolic BP range: 0 - 299; Heart rate range: 40 - 180. These values represent the reliable ranges for the device. For each variable, higher values are generally considered "worse" and lower values "better." However, very low values (e.g., systolic BP values <80, diastolic BP values <60, and HR values <50) may also indicate poor cardiovascular health.
Hypnotic Use | 9 weeks, 6 months, 12 months
  Daily hypnotic use is self-reported in a 7-day sleep diary, with the ability to report up to 3 medications taken on a given night.
  Scale Range: 22 Minimum Score: 0 (no hypnotic medication use on any day; better) Maximum Score: 21 (multiple hypnotic medications and/or multiple days of use; worse).
  Retrospective hypnotic use in past 3 months is self-reported in a demographic and health care utilization questionnaire.
  Scale Range: 0 - no limit Minimum Score: 0 (better) Maximum Score: no limit (multiple hypnotic medications and/or multiple days of use; worse).
Health Care Utilization | 9 weeks, 6 months, 12 months
  The Health care utilization Questionnaire is a self-report measure that asks about recent health care services that have been sought and medications for hypertension and insomnia.
  Scale Range: 0 - no limit Minimum Score: 0 (no visits or medications; better) Maximum Score: no limit (multiple visits and/or medications; worse)
Health-Related Quality of Life | 9 weeks, 6 months, 12 months
  The Rand-12 is a 12-item self-report measure that produces physical health (PHC) and mental health (MHC) component scores. T-scores are used and have a population mean of 50.
  Scale Range (PHC and MHC): 100 Minimum Score (PHC and MHC) = 0 (worse) Maximum Score (PHC and MHC) = 100 (better)
Client Satisfaction | 9 weeks
  The Client Satisfaction Questionnaire (CSQ) is an 8-item self-report measure that assesses client satisfaction with the services they received.
  Scale Range: 24 Minimum Score = 8 (low satisfaction) Maximum Score = 32 (high satisfaction)
Provider Satisfaction | Following closing of recruitment
  The provider satisfaction questionnaire is a self-report measure that assesses provider's perceived efficacy of the treatments their patients received, barriers to treatment, and satisfaction of both providers and patients.
  Scale Range: 38 Minimum Score: 0 (low satisfaction) Maximum Score: 37 (high satisfaction)

OTHER OUTCOMES:
Daytime Impairment Related to Sleep | 9 weeks, 6 months, 12 months
  PROMIS Sleep Related Impairment is a self-report measure that assesses problems related to insufficient sleep during the past 7 days. It is administered by computerized adaptive testing (CAT) with individual responses guiding the system's choice of subsequent items from the full 16-item bank.
  Scale Range: Item responses are combined to yield a T-score with population mean of 50, standard deviation of 10, and range of ~20 - ~80. Higher scores indicate greater sleep related impairment.
Side Effects | 9 weeks, 6 months, 12 months
  Side effects (frequency, severity, impairment) are recorded via a self-report that was adapted from the Fisber.
  Range: 22 Minimum Score: 0 (no side effects; better) Maximum Score: 21 (worse)
  Those reporting severity of > moderate and/or frequency > 50% of the time in their self-report, or who spontaneously report a side effect, are contacted by the study coordinator. Information is gathered regarding the nature and duration of the event and action taken. Determination of causality and outcomes attributed to the event are then made.
Insomnia Severity | 9 weeks, 6 months, 12 months
  The Insomnia Severity Index (ISI) is a 7-item self-report questionnaire that measures severity of insomnia symptoms during the last two weeks.
  Scale Range: Minimum Score = 0 (no insomnia); Maximum Score = 28 (severe insomnia)
Sleep Quality | 9 weeks, 6 months, 12 months
  The Pittsburgh Sleep Quality Index (PSQI) is an 18-item self-report measure that assesses sleep quality in the past month. These items are combined into seven component scores (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medication, and daytime dysfunction). The seven component scores are added to produce a global sleep quality score. Higher global scores reflect lower sleep quality, with 5 as a cut-off distinguishing good from poor sleepers.
  Scale Range: 22
  Minimum Score = 0 (better); Maximum Score = 21 (worse)
Daytime Sleepiness | 9 weeks, 6 months, 12 months
  The Epworth Sleepiness Scale (ESS) is an 8-item self-report measure that assesses daytime sleepiness by asking about the likelihood of dozing in certain situations. Individual items are summed to yield the ESS score.
  Scale Range: 25
  Minimum Score = 0 (never doze); Maximum Score = 24 (doze a lot)
Falls | 9 weeks, 6 months, 12 months
  Falls are recorded via self-report.
  Range: 5 Minimum Score: 0 (no falls; better) Maximum Score: 5 (> 4 falls; worse)
  Those reporting a fall are contacted by the coordinator and information is gathered regarding the date and time of day of the fall(s), proximity to a sleep episode, contributing factors, and whether or not medication for sleep or anxiety were taken in the 24 hours preceding the fall.
Improvement | 9 weeks, 6 months, 12 months
  The Patient Global Impression of Improvement (PGI-I) Scale is a self-report measure that rates perceived response to intervention.
  Scale Range: 7 Minimum Score: 1 (very much improved; better) Maximum Score: 7 (very much worse; worse)
Bed times | Intervention, 9 weeks, 6 months, 12 months
  The in and out of bed times are recorded in a 7-day sleep diary and include: bed time, lights out time, wake time, and out-of-bed time. Bed time is the clock time when the participant got into bed. Lights out time is the clock time when the participant actually attempted to sleep (i.e., turned out the lights). Wake time is the clock time of the participant's final awakening. Out-of-bed time is the clock time they got out of bed for the day.
  Ranges for these clock-time variables use 24 hours, with no minimum or maximum value.
Time to fall asleep | Intervention, 9 weeks, 6 months, 12 months
  Time to fall asleep is recorded in a 7-day sleep diary.
  Range: 24 hours Minimum value = 0 minutes (better) Maximum value = 1440 minutes (worse)
Wake After Sleep Onset (WASO) | Intervention, 9 weeks, 6 months, 12 months
  WASO is recorded in a 7-day sleep diary, and refers to the number of minutes of wakefulness between the time of falling asleep and Wake Time.
  Range: 24 hours Minimum value = 0 minutes (better) Maximum value = 1440 minutes (worse)
Subjective Sleep Quality | Intervention, 9 weeks, 6 months, 12 months
  Subjective sleep quality is recorded in a 7-day sleep diary.
  Range: 5 Minimum score: 0 (very poor; worse) Maximum score: 4 (very good; better)
Use of Sleep Medication | Intervention, 9 weeks, 6 months, 12 months
  Use of sleep medication is recorded in a 7-day sleep diary, with the ability to report up to 3 medications taken on a given night.
  Scale Range: 22
  Minimum Score: 0 (no sleep medication use on any night; better) Maximum Score: 21 (multiple sleep medications and/or multiple nights of use; worse).
Sleep Efficiency | Intervention, 9 weeks, 6 months, 12 months
  Sleep Efficiency is calculated from values recorded in a 7-day sleep diary. It refers to the percentage of time asleep while in bed. Time in bed is calculated as (Out of bed time) - (Bed time), in minutes. Sleep efficiency is calculated as (Total sleep time/time in bed) X 100.
  Range: 101 Minimum for sleep efficiency: 0% (worse) Maximum for sleep efficiency: 100% (better)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Buysse, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Health System, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make available to the research community any resource that is presented in a publication that is published or accepted for publication. We agree to release and share data in a timely manner, but no later than one year following completion of the funded project period or the date of publication of the main findings from our final data set.
  Data will be provided in the form of an Access data base.
  A data dictionary will be provided to define all data fields.
  We will not provide data analytic tools.
  We are providing this Data Sharing Agreement in keeping with the requirements of RFA-HL-14-019.
  Data will be shared as Access data base(s), provided in electronic format by e-mail or durable media.
Time Frame: We agree to release and share data in a timely manner, but no later than one year following completion of the funded project period or the date of publication of the main findings from our final data set.
Access Criteria: We will share data with investigators working at an institution with a Federal Wide Assurance.
  To gain access to data, researchers must submit a detailed description of their project. The proposal must include the investigator's personal identification and institutional affiliation, a current CV, qualifications, estimated duration of the proposed research, source of financial support, and a conflict of interest statement. The protocol described must include study aims, background and significance, and methods and types of analysis, and a description of the data requested and list of variables. Once approved, the investigator must complete the necessary University of Pittsburgh IRB exempt research application form and document completion of a responsible conduct of research program. Data will be prepared by an 'honest broker.' Data will not be provided that could identify individual research participants or that the original consent form expressly forbade.

REFERENCES:
- [Derived] Levenson JC, Rollman BL, Ritterband LM, Strollo PJ, Smith KJ, Yabes JG, Moore CG, Harvey AG, Buysse DJ. Hypertension with unsatisfactory sleep health (HUSH): study protocol for a randomized controlled trial. Trials. 2017 Jun 6;18(1):256. doi: 10.1186/s13063-017-2001-9. PMID 28587609

DOCUMENTS (1):
  • Informed Consent Form (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/29/NCT02508129/ICF_000.pdf